CLINICAL TRIAL: NCT02610959
Title: Iodine Status During Pregnancy and Its Effect on Infant Development; a Randomized Intervention Study With Cod
Brief Title: Iodine Status During Pregnancy and Its Effect on Infant Development.
Acronym: Mommy'sFood
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Nutrition and Seafood Research, Norway (Other Government)
Collaborators: NORCE Norwegian Research Centre AS (Other)
Responsible Party: Principal Investigator, Marian Kjellevold, PhD, Scientist, National Institute of Nutrition and Seafood Research, Norway
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2015/879
Record Dates: First submitted 2015-11-17; First posted 2015-11-20 (Estimated); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Diet; Neurodevelopment
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention group (Experimental): Intervention with cod 200 grams two times the week for four months.
  Interventions: Other: Intervention group
- Control group (Experimental): Control group which will continue to eat their habitual diet.
  Interventions: Other: Control group

INTERVENTIONS:
Other: Intervention group — The overall aim of the present project is to investigate if intake of cod in pregnancy has impact on infant development up to 12 month.
  Arms: Intervention group
Other: Control group — The overall aim of the present project is to investigate if intake of cod in pregnancy has impact on infant development up to 12 month.
  Arms: Control group

SUMMARY:
The overall aim of the present project is to investigate if intake of cod in pregnancy has impact on infant development up to 12 month. 142 pregnant women will be allocated into two groups, one counsuming cod two times the week for four months and one group will continue to follow their habitual diet. To study this, urine samples, dietary data and blood samples from the mother and from the infant, as well as data on neurodevelopment and cognitive functioning will be collected at several time points.

DETAILED DESCRIPTION:
The World Health Organization considers iodine deficiency to be "the single most important preventable cause of brain damage" worldwide. The effect of severe iodine deficiency is well documented. Pregnant and nursing mothers have increased requirements and are thus a vulnerable group. Iodine is a key component of thyroid hormones that are critical for normal development of the brain and nervous system in utero. There is little data on the effect of mild- and moderate iodine deficiency. Results from the Norwegian Mother and Child cohort (n = about 62,000) shows that only 22% of the participants had an iodine intake, estimated from food frequency questionnaire, that meets the recommendations of WHO / UNICEF / ICCIDD. Urine samples from a sub-sample (n = 119) confirmed suboptimal iodine status. The results are consistent with recent data from a NIFES study of about 100 women from the municipality of Fjell, which reviled suboptimal iodine status both in pregnancy and three months after birth. Preliminary results from the study Little in Norway, where NIFES measured the iodine status in approximately 1,000 pregnant from across the country, is also consistent with these investigations. Dairy products is highlighted as the main source of iodine for the participants in the Norwegian Mother and Child cohort, while lean fish is the food group that has the highest Iodine levels. In this article, the positive effect of seafood was explained by the fatty acids EPA and DHA, while the latest publication suggests that the effect of an adequate intake of seafood during pregnancy are more complex, and that the high iodine levels in seafood may also be important. Based on this knowledge, there is a need for an intervention study where pregnant consume cod regularly over a longer period and where the children are followed up over time. Thus, in the present project the researchers will investigate if intake of cod in pregnancy has impact on infant development up to 12 month. 142 pregnant women will be allocated into two groups, one consuming cod two times the week for four months and one group will eat as normal. Urine samples, dietary data and blood samples from the mother and from the infant, as well as data on neurodevelopment and cognitive functioning will be collected at several time points.

ELIGIBILITY:
Inclusion Criteria:

* ≤ gestational week 19,
* prim parous,
* singleton pregnancy,
* Norwegian speaking and / or understand Norwegian writing due to all validated tests of the child will be in Norwegian.

Exclusion Criteria:

* allergies to fish,
* chronic diseases known to affect iodine status (Graves' disease, Thyroiditis, Thyroid Nodules, known hypothyroidism, known hyperthyroidism).

Ages: 16 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 137 (Actual)
Dates: Start 2015-12; Primary Completion 2018-09-01 (Actual); Study Completion 2018-09-17 (Actual)

PRIMARY OUTCOMES:
Difference in Urinary iodine concentration between groups | 16 weeks
  A collection sample of 1 ml of homogenized spot morning urin collected on six consecutive days will be analyzed for iodine (umol/L) before and after the intervention in both Groups. Groups will be compared in relation to delta-values before and after intervention/no intervention.

SECONDARY OUTCOMES:
Difference in Bayley Scale of Infant Developmental scores between groups | 17 months
  Student's t-test to compare the means between the groups.

OTHER OUTCOMES:
Difference in Ages and Stages Questionnaire: Social-Emotional (ASQ:SE) | Infant age 3, 6 and 11 months
  We compare scores between groups using linear mixed effects models and examined whether iodine status post intervention mediated the effect on child development.
Difference in Ages and Stages Questionnaire 2nd. edition (ASQ-2) | Infant age 3, 6 and 11 months
  We compare scores between groups using linear mixed effects models and examined whether iodine status post intervention mediated the effect on child development.
Extended follow up at five-six years - 5-15R (FTF/Five To Fifteen) questionnaire | Child age five-six years
  We compare scores between groups 5-15R (FTF/Five To Fifteen) questionnaire
Extended follow up at five-six years - Difference in Ages and Stages Questionnaire Social-Emotional (ASQ:SE) | Child age five-six years
  We compare scores between groups in Ages and Stages Questionnaire: Social-Emotional (ASQ:SE)
Extended follow up at five-six years - Strengths and Difficulties Questionnaire | Child age five-six years
  We compare scores between groups in Strengths and Difficulties Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Marian Kjellevold, PhD, Study Chair — Institute of Marine Research
Locations (1):
- Institute of Marine Research, Bergen, Norway

REFERENCES:
- [Derived] G Bjorkevoll SM, Konijnenberg C, Kvestad I, McCann A, Ueland PM, Naess Sleire S, Dahl L, Kjellevold M, Strand TA, Markhus MW. Vitamin B12 and Folate Status in Pregnant Females and Their Infants in Norway: Secondary Analysis from the Mommy's Food Study. J Nutr. 2023 Dec;153(12):3543-3554. doi: 10.1016/j.tjnut.2023.10.013. Epub 2023 Oct 18. PMID 37858724
- [Derived] Naess S, Markhus MW, Strand TA, Kjellevold M, Dahl L, Stokland AM, Nedrebo BG, Aakre I. Iodine Nutrition and Iodine Supplement Initiation in Association with Thyroid Function in Mildly-to-Moderately Iodine-Deficient Pregnant and Postpartum Women. J Nutr. 2021 Oct 1;151(10):3187-3196. doi: 10.1093/jn/nxab224. PMID 34255063
- [Derived] Kvestad I, Hysing M, Kjellevold M, Naess S, Dahl L, Markhus MW. Maternal Cod Intake during Pregnancy and Infant Development in the First Year of Life: Secondary Analyses from a Randomized Controlled Trial. J Nutr. 2021 Jul 1;151(7):1879-1885. doi: 10.1093/jn/nxab083. PMID 33847344
- [Derived] Markhus MW, Hysing M, Midtbo LK, Nerhus I, Naess S, Aakre I, Kvestad I, Dahl L, Kjellevold M. Effects of Two Weekly Servings of Cod for 16 Weeks in Pregnancy on Maternal Iodine Status and Infant Neurodevelopment: Mommy's Food, a Randomized-Controlled Trial. Thyroid. 2021 Feb;31(2):288-298. doi: 10.1089/thy.2020.0115. Epub 2020 Sep 8. PMID 32746774
- [Derived] Naess S, Kjellevold M, Dahl L, Nerhus I, Midtbo LK, Bank MS, Rasinger JD, Markhus MW. Effects of seafood consumption on mercury exposure in Norwegian pregnant women: A randomized controlled trial. Environ Int. 2020 Aug;141:105759. doi: 10.1016/j.envint.2020.105759. Epub 2020 May 7. PMID 32388274
- [Derived] Markhus MW, Kvestad I, Midtbo LK, Nerhus I, Odegaard ER, Graff IE, Lie O, Dahl L, Hysing M, Kjellevold M. Effects of cod intake in pregnancy on iodine nutrition and infant development: study protocol for Mommy's Food - a randomized controlled trial. BMC Nutr. 2018 Feb 17;4:7. doi: 10.1186/s40795-018-0215-1. eCollection 2018. PMID 32153871
- [Derived] Naess S, Aakre I, Kjellevold M, Dahl L, Nerhus I, Midtbo LK, Markhus MW. Validation and reproducibility of a new iodine specific food frequency questionnaire for assessing iodine intake in Norwegian pregnant women. Nutr J. 2019 Oct 29;18(1):62. doi: 10.1186/s12937-019-0489-4. PMID 31665021